# **PROVESA** trial

Proficiency based progression training for robotic vesico-urethral anastomosis chicken model versus the Halsted's model: a cross-specialty, multicentric, randomized and blinded clinical trial.

## **Study Protocol**

Principal Investigator: Ruben De Groote, MD

Research center: ORSI Academy, Melle, Belgium

July 27th 2020

NCT ID not yet assigned

Ethical Committee approval number 22072020

## **Summary**

In a prospective, randomized and blinded study robotic naïve (urology (n = 12), surgery (n = 12) and gynecology (n = 12)) residents (n = 36) from the KU Leuven and University of Gent residency training programs will be randomized (in equal discipline numbers) to Traditional Halstedian apprenticeship type training or proficiency based progression (PBP) training to learn to perform a vesico-urethral anastomosis (VUA) on a chicken model. Both groups will receive the same e-learning (on how to perform the VUA on the chicken model) and skills laboratory robotic training curriculum. The PBP trained group will however be required to demonstrate quantitively defined proficiency benchmarks for training progression (i.e., from e-learning to the skills lab). The PBP group will also have a defined benchmark to demonstrate before training is deemed completed. The Traditional trained group will train in the same skills laboratory for a case-matched period of time as the PBP group, with the same level of supervising faculty proctors and using the same training resources but with no proficiency benchmarks or metric-based feedback. Both groups will be required to perform a VUA on the chicken model before skills training proper and at the end of training. Investigators will be trained in pairs to assess VUA performance from a pre-defined set of explicitly defined binary metric events reliably (inter-rater reliability > 0.8). They will also be blinded as to the identity of the trainee performing the procedure, how they were trained (i.e., group) and procedure order.

H<sub>1</sub> It is hypothesisied that iimplementation of PBP training in teaching the robotic suturing of VUA leads to better surgical training outcomes (i.e., lower number of performance errors) when compared to Halsted's method.

Proficiency based progression training for robotic vesico-urethral anastomosis chicken model versus the Halsted's model: a prospective, randomized and blinded clinical trial.

#### Introduction

Current surgical training is outdated.<sup>1</sup> The Halsted's model 'See one, Do one, Teach one', is still widely used during training of surgeons. Consequently, a patient is still exposed to a novice resident who does the procedure for the very first time. For too long, surgical training is dependent on the quality of the trainer with a lack of systematics, standardization and objective scoring systems.<sup>2</sup> Because of financial and ethical reasons, it can no longer be justified that the beginning of a learning curve takes place in the operating room on real life patients. By mitigating the initial learning curve in an out-of-hospital setting and by developing a standardized, novel training system, patient safety could be improved.

Proficiency Based Progression (PBP)<sup>3-5</sup> training or Quality Assured Training is a novel training method that already has demonstrated its value in different surgical specialties.<sup>6-12</sup> In this kind of training a specific level of performance defined by a quantitative score (benchmark) or scores on a standardized assessment must be demonstrated to gain the proficiency level. Only demonstrating the ability to meet quantitatively defined performance benchmarks permits progression in training (i.e., proficiency-based progression [PBP] training).

## **Background**

Suturing and knot tying are fundamental skills for all surgical disciplines. They serve an important clinical function but using a minimally invasive approach means that they are even more challenging to complete. A curricular approach to learning laparoscopic suturing and knot tying has been successfully demonstrated for Nissen fundoplication.<sup>10</sup>

Fundamental in creating a proficient robotic surgeon is the acquisition of basic surgical skills, such as suturing and knot tying. Some training models mimic the real anatomical environment in which a procedure will be performed and provide trainees with the opportunity to learn and practice their skills before starting their practice on real cases in the operating room. Numerous dry-lab, wet-lab, and virtual reality simulation models have been described. The "Venezuelan chicken model" is generally accepted as a optimal model for trainees to learn robotic suturing, anastomosis and knot tying tasks (for all surgical disciplines). We will use the Venezuelan chicken model in this study. It has several advantages; it is inexpensive, widely available, easy to prepare, it is a good model for the urethro-vesical anastomosis training, it is possible to introduce a catheter and performing the leakage test, it takes the trainee approx. 20 mins to complete the task. Over the past 12 months ORSI has developed and validated (Delphi consensus and Construct Validity) performance metrics for the task.

This study aims to compare the effectiveness of Halsted's apprenticeship approach to training with the Proficiency Based Progression (PBP) approach for teaching the robotic suturing of a vesico-urethral anastomosis (VUA) on a chicken model.

#### Methods

#### **Subjects**

Robotic naïve urology (n = 12), surgery (n = 12) and gynecology (n = 12) residents (n = 36) from the UKU Leuven and University of Gent residency training programs will participate. They will be randomized (using an online randomizer <a href="https://www.random.org/">https://www.random.org/</a>) to teaching of VUA suturing with either Halsted's (n = 18) or the PBP method including procedure-specific, validated metrics (n = 18).

## Procedure and training

Trainees in the Traditional trained group will be trained according to the traditional approach of 'See one, do one, teach one' principle. Trainees will have a e-learning didactic component (specifically on the anatomy & physiology of the procedure, clinical aspects of the procedure, published evidence etc) which they must complete before training by a procedure expert. On completion of the e-learning module they will complete a summative assessment of their knowledge. They will then be shown how and then trained to suture and tie knots using the robot. The VUA will be demonstrated initially by an expert and who will then proctor the trainees in the same technique for repeated training trials., i.e., repeated practice for a period of time matched to the PBP group.

Students in the PBP trained group will follow the exact same e-learning didactic course as the Traditional trained group but the PBP group will be required to pass a test of procedure knowledge before continuing to the surgical training. Their knowledge will be assessed in a formative and summative fashion. After their initial VUA assessment, procedure-specific and validated procedure metrics will be used to teach the students the steps of the procedure, as well as the correct (and incorrect) way to perform the procedure. The metrics will be used to give them performance feedback with specific advice on how they might improve their performance, i.e., deliberate practice.<sup>17</sup>

Both groups of subjects will receive the exact same amount of training and have access the same didactic and training resources. Both groups will also complete a baseline assessment on the chicken model before technical skills training. Assessors, blinded to group membership and procedure order (first or last procedure) will evaluate each student's first and final VUA with the validated chicken anastomosis metrics. They will also assess performance with the GEARS<sup>18</sup> assessment tool (Figure 2). Additionally, the student's satisfaction of the training method will be assessed using a Likert scale 1-5 (Figure 3).

Proficiency Definition: In the study proposed here proficiency levels will be quantified and defined on the objectively assessed performance of surgeons experienced in performing that VUA task being trained. This performance level will be established from the construct validation study of the procedure metrics derived from the procedure characterizations.<sup>4, 5, 19</sup>

#### Performance assessments

Investigators will be trained in pairs to assess performance from a pre-defined set of explicitly defined metric events reliably (inter-rater reliability > 0.8). They will be blinded as to the identity of the trainee performing the procedure, how they were trained (i.e., group) and procedure order.

#### **Procedure performance assessment**

We will record how long subjects took to perform the procedure, the number of steps correctly completed and procedure errors/deviations from optimal performance. We will also record and cost the instrumentation/needles/suture etc utilised in the performance of the procedure.

**Baseline Assessment**: -Prior to the commencement of education and training protocol all subjects from both groups will be assessed on their performance of the VUA task. Performance on the procedure will be video recorded and assessed as previously described.

**Statistical Analysis**: From previous similar studies, it has been found that data has been reasonably normally distributed and suitable for parametric statistical analysis. If the data violates any of the assumptions of normality, data will be compared for statistical significance with Mann-Whitney U for comparison between two independent samples and Wilcoxon signed-rank test. Where data are normally distributed with approximately equal variance differences between groups, task performance will be compared for statistical significance with two-factor Analysis of Variance where factor one is the type of training subjects received and factor two is the order the task was performed (i.e, baseline

performance and end of training performance). The same analysis will be used to assess the binary checklist metric scores and the GEARS scores (seperatly) for the Standard trained and the PBP trained groups. Specific post hoc statistical contrasts between surgeon groups performance within a training condition (i.e., between the objectively assessed performance of urology, surgery and gynecology residents) will be done with Scheffe F-tests.

**Statistical power calculation**: A pilot study has shown that novices on average make 16.6 (SD = 4) performance errors on the task. Assuming a reduction of  $\sim$ 40% with PBP training (i.e., 16.6 vs 10 errors) with a standard deviation of n = 4, an Alpha – 1% with 16 subjects in each group would yield a statistical power of 0.998 for the proposed study.



- \* By assessors blinded to group membership and procedure order (first or last procedure)
- \*\* Matching according to specialty

**Figure 1**. the design of the prospective randomized study to evaluate the impact of PBP on learning the robotic surgical skills for a vesico-urethral anastomis (VUA) on a chicken model.

#### Hypothesis

- H<sub>1</sub> Implementation of PBP training in teaching the robotic suturing of VUA leads to better surgical training outcomes (i.e., lower number of performance errors) when compared to Halsted's method.
- H<sub>0</sub> There will be no difference in the procedure knowledge prior to VUA training
- H<sub>0</sub> There will be <u>no</u> difference in the objectively assessed procedure performance of the urology, surgery and gynecology residents at the end of training in the PBP group
- H<sub>0</sub> There <u>will</u> be a difference in the objectively assessed procedure performance of the urology, surgery and gynecology residents at the end of training in the Traditional trained groups.
- H<sub>0</sub> There will be no difference in student satisfaction with the two approaches to training.

| 1 | 2 | 3 | 4 | 5 |
|---|---|---|---|---|
| Constantly overshoots | | Some overshooting or | | Accurately directs |
| target, wide swings, | | missing of target, but | | instruments in the |
| slow to correct | | guick to correct | | correct plane to target |
| | | 4 | | con out plante to tanget |
| Bimanual dexterity | | | | |
| 1 | 2 | 3 4 | | 5 |
| Uses only one hand, | | Uses both hands, but | | Expertly uses both |
| ignores nondominant | | does not optimize | | hands in a |
| hand, poor coordination | | interaction between | | complementary way to |
| | | hands | | provide best exposure |
| Efficiency | | | | |
| í | 2 | 3 | 4 | 5 |
| Inefficient efforts; | | Slow, but planned | | Confident, efficient and |
| many uncertain | | movements are | | safe conduct, maintains |
| movements; constantly | | reasonably organized | | focus on task, fluid |
| changing focus or | | | | progression |
| persisting without | | | | |
| progress | | | | |
| Force sensitivity | | | | |
| 1 | 2 | 3 | 4 | 5 |
| Rough moves, tears | | Handles tissues | | Applies appropriate |
| tissue, injures nearby | | reasonably well, minor | | tension, negligible |
| structures, poor | | trauma to adjacent | | injury to adjacent |
| control, frequent | | tissue, rare suture | | structures, no suture |
| suture breakage | | breakage | | breakage |
| Autonomy | | | | |
| 1 | 2 | 3 | 4 | 5 |
| Unable to complete | | Able to complete task | | Able to complete task |
| entire task, even with | | safely with moderate | | independently without |
| verbal guidance | | guidance | | prompting |
| Robotic control | | | | |
| 1 | 2 | 3 | 4 | 5 |
| Consistently does not | | View is sometimes not | | Controls camera and |
| optimize view, hand | | optimal. Occasionally | | hand position optimally |
| position, or repeated | | needs to relocate | | and independently. |
| collisions even with | | arms. Occasional | | Minimal collisions or |
| guidance | | collisions and | | obstruction of assistant |
| guidance | | | | |
| guidance | | obstruction of assistant. | | |

Figures 2. The GEARS assessment tool

## TRAINING EVALUATION FORM

Disagree

Disagree

Disagree

Neutral

Neutral

Neutral

Agree

Agree

Agree

| Instructor: Date: | ( | (Please fill out one for each instructor) | | | |
|---|---|---|---|---|---|
| Training Quality | · | 22 | Đ); | 22 | 500 |
| The overall quality of the training I received was high | Strongly<br>Disagree | Disagree | Neutral | Agree | Strongly<br>Agree |
| This training will be beneficial to me<br>in the performance of my job | Strongly<br>Disagree | Disagree | Neutral | Agree | Strongly<br>Agree |
| Course Presentation | | | | | |

Strongly Disagree

Strongly

Disagree

Strongly

Disagree

| The vocabulary used in the course<br>was clear and easy to understand. | Strongly<br>Disagree<br>Strongly<br>Disagree | Disagree<br>Disagree | Neutral<br>Neutral | Agree<br>Agree | Strongly<br>Agree<br>Strongly<br>Agree |
|---|---|---|---|---|---|
| The instructor was knowledgeable<br>and effective. | | | | | |
| Course Objectives | | | | | |
| The course covered the material I expected. | Strongly<br>Disagree | Disagree | Neutral | Agree | Strongly<br>Agree |
| The times scheduled for the agenda<br>items were appropriate. | Strongly<br>Disagree | Disagree | Neutral | Agree | Strongly<br>Agree |
| The course met the training objectives. | Strongly<br>Disagree | Disagree | Neutral | Agree | Strongly<br>Agree |
| The course met my training needs. | Strongly<br>Disagree | Disagree | Neutral | Agree | Strongly<br>Agree |

Figure 3: Likert-scale for the assessment of training satisfaction

The methods of content delivery

The topics were presented in a

appropriate for this course.

The course material was easy to

understand and helpful.

logical order.

(lectures, PowerPoints, etc.) were

Strongly Agree

Strongly

Agree

Strongly

Agree

#### References

- 1. Pellegrini CA. Surgical education in the United States: navigating the white waters. *Annals of Surgery* 2006; 244(3):335 342.
- 2. Cuschieri A. Whither minimal access surgery: tribulations and expectations. *The American Journal of Surgery* 1995; 169(1):9 19.
- 3. Gallagher A. Metric-based simulation training to proficiency in medical education:-What it is and how to do it. *Ulster Medical Journal* 2012; 81(3):107-113.
- 4. Gallagher AG, O'Sullivan GC. Fundamentals of Surgical Simulation; Principles & Practices London: Springer Verlag, 2011.
- 5. Gallagher AG, Ritter EM, Champion H, et al. Virtual reality simulation for the operating room: proficiency-based training as a paradigm shift in surgical skills training. *Annals of surgery* 2005; 241(2):364-372.
- 6. Breen D, O'Brien S, McCarthy N, et al. Effect of a proficiency-based progression simulation programme on clinical communication for the deteriorating patient: a randomised controlled trial. *BMJ open* 2019; 9(7):e025992.
- 7. Srinivasan KK, Gallagher A, O'Brien N, et al. Proficiency-based progression training: an 'end to end'model for decreasing error applied to achievement of effective epidural analgesia during labour: a randomised control study. *BMJ open* 2018; 8(10):e020099.
- 8. Cates CU, Lönn L, Gallagher AG. Prospective, randomised and blinded comparison of proficiency-based progression full-physics virtual reality simulator training versus invasive vascular experience for learning carotid artery angiography by very experienced operators. *BMJ Simulation and Technology Enhanced Learning* 2016; 2(1):1-5.
- 9. Angelo RL, Ryu RK, Pedowitz RA, et al. A proficiency-based progression training curriculum coupled with a model simulator results in the acquisition of a superior arthroscopic Bankart skill set. *Arthroscopy: The Journal of Arthroscopic & Related Surgery* 2015; 31(10):1854-1871.
- 10. Van Sickle K, Ritter EM, Baghai M, et al. Prospective, randomized, double-blind trial of curriculum-based training for intracorporeal suturing and knot tying. *Journal of the American College of Surgeons* 2008; 207(4):560-8.
- 11. Ahlberg G, Enochsson L, Gallagher AG, et al. Proficiency-based virtual reality training significantly reduces the error rate for residents during their first 10 laparoscopic cholecystectomies. *The American Journal of Surgery* 2007; 193(6):797-804.
- 12. Seymour NE, Gallagher AG, Roman SA, et al. Virtual reality training improves operating room performance: results of a randomized, double-blinded study. *Annals of Surgery* 2002; 236(4):458-63; discussion 463-4.
- 13. Vanlander AE, Mazzone E, Collins JW, et al. Orsi Consensus Meeting on European Robotic Training (OCERT): Results from the First Multispecialty Consensus Meeting on Training in Robot-assisted Surgery. *Eur Urol* 2020.
- 14. Cacciamani G, De Marco V, Siracusano S, et al. A new training model for robotassisted urethrovesical anastomosis and posterior muscle-fascial reconstruction: the Verona training technique. *J Robot Surg* 2017; 11(2):123-128.
- 15. Santos DRD, Calvo FC, Feijo DH, et al. New training model using chickens intestine for pediatric intestinal anastomosis. *Acta Cir Bras* 2019; 34(7):e201900709.
- 16. Sotelo RJ, Astigueta JC, Carmona OJ, et al. Chicken gizzard: a new training model for laparoscopic urethrovesical anastomosis. *Actas Urol Esp* 2009; 33(10):1083-7.

- 17. Ericsson KA, Krampe RT, Tesch-Römer C. The role of deliberate practice in the acquisition of expert performance. *Psychological Review* 1993; 100(3):363-406.
- 18. Goh AC, Goldfarb DW, Sander JC, et al. Global evaluative assessment of robotic skills: validation of a clinical assessment tool to measure robotic surgical skills. *The Journal of urology* 2012; 187(1):247-252.
- 19. Gallagher AG, Ritter EM, Satava RM. Fundamental principles of validation, and reliability: rigorous science for the assessment of surgical education and training. *Surgical Endoscopy* 2003; 17(10):1525-9.